CLINICAL TRIAL: NCT03760523
Title: Phase 1/1b Dose Escalation Study of Minnelide in Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Dose Escalation Study of Minnelide in Relapsed or Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Toxicity -Two DLT events occurred
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Minneamrita Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19742
Record Dates: First submitted 2018-11-27; First posted 2018-11-30 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: leukemia; myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia; Leukemia, Myeloid | interventions — 14-O-phosphonooxymethyltriptolide disodium salt

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Minnelide Dose Escalation (Experimental): A 3+3 design will be used. The first 3 patients will be treated at dose level 1. If none experience a Dose Limiting Toxicity (DLT), the next 3 patients will be treated at dose level 2. If a DLT is observed in 1 out of 3 patients at dose level 1, up to an 3 more patients will be enrolled and treated at that dose level. If 2 patients at dose level have DLTs, dosing will be lowered to dose level -1 (.5 mg daily, taken orally). If 2 or more of the up to 6 patients at any dose level have DLTs, the preceding dose will be declared the Maximum Tolerated Dose (MTD). If more than 1 DLT occurs at Dose Level -1, the investigators will consider stopping the study. Once the MTD has been established, an additional 10 patients will be enrolled at this level to better characterize safety and tolerability.
  Interventions: Drug: Minnelide

INTERVENTIONS:
Drug: Minnelide — Patients will take Minnelide orally once daily on Days 1-21 of 28 day Cycle. Dose Escalation Schedule: Dose Level -1: .5 mg, Dose Level 1: .75 mg, Dose Level 2: 1 mg, Dose Level 3: 1.25 mg.

SUMMARY:
This study is to determine the safety and recommended dosing of Minnelide in Acute Myeloid Leukemia (AML)

DETAILED DESCRIPTION:
This phase 1 dose escalation clinical trial will establish the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of Minnelide as single-agent in relapsed/refractory (R/R) acute myeloid leukemia (AML) patients who are ineligible to receive intensive chemotherapy. The oral formulation of Minnelide will be used. Minnelide is a prodrug of triptolide (a potent heat shock protein (HSP) 70 inhibitor) with promising preclinical activity in AML.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18 years or older.
* Participant must have relapsed or refractory acute myeloid leukemia (AML) (excluding acute promyelocytic leukemia).
* Relapsed patients must have received at least 1 induction chemotherapy regimen or two cycles of a hypomethylating agent and achieved a Complete Response (CR), followed by relapse of disease.
* Refractory patients must have received at least 1 induction chemotherapy regimen or two cycles of hypomethylating agent without achieving a CR.
* Eastern Cooperative Oncology Group (ECOG) performance status <2.
* Participants must have acceptable organ function.
* Be able and willing to adhere to the study visit schedule and other protocol requirements.
* Must be able to swallow capsules and have no evidence of GI tract abnormality that would alter the absorption of oral medications.
* The effects of Minnelide on the developing human fetus are unknown. For this reason, women of child-bearing potential must have a negative serum or urine pregnancy test within 24 hours prior to beginning study treatment.
* Participants of childbearing potential must practice contraception. Females of childbearing potential: Recommendation is for 2 effective contraceptive methods during the study. Male participants with female partners who are of childbearing potential: Recommendation is for male and partner to use at least 2 effective contraceptive methods, as described above, during the study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Minnelide, breastfeeding mothers must agree to discontinue nursing if the mother is treated with Minnelide.
* Provision of signed and dated informed consent document
* Patients with prior allogeneic stem cell transplant who experience relapse of AML are eligible if they are off of immunosuppressive therapy and without any evidence of graft-versus-host disease (GVHD)

Exclusion Criteria:

* Participants may not have received any therapy with any investigational products, systemic anti-neoplastic therapy, or radiotherapy within 14 days prior to Cycle 1 Day 1. Patients actively receiving hydroxyurea are eligible and may continue to receive hydroxyurea during protocol treatment.
* Candidates for standard and/or potentially curative treatments.
* Major surgery within 28 days prior to Cycle 1 Day 1.
* New York Heart Association Class III or IV heart failure, myocardial infarction within the past 6 months, unstable arrhythmia, or evidence of ischemia on an electrocardiogram (EKG)
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* Known, active HIV, Hepatitis A, B or C infection (prior Hepatitis C infection that has been treated and determined to be cured is allowed)
* Symptomatic central nervous system (CNS) involvement with leukemia
* A concurrent second active and non-stable malignancy with the exception of non-melanoma skin cancer or carcinoma in-situ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2023-10-09 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Minnelide | Up to 28 days for each dosing cohort
  MTD will be determined by testing increasing doses up to 1.25 mg daily. MTD reflects highest dose of drug that did not cause a Dose Limiting Toxicity (DLT).
Number of Participants Who Experience Dose Limiting Toxicities (DLTs) | Up to 28 days for each dosing cohort
  A DLT is any Grade 3 or 4 drug-related non-hematologic toxicity, with some exceptions per protocol.

SECONDARY OUTCOMES:
Complete Response (CR) | Up to 12 months
  Participants who experience Complete Response (CR) and Complete Response with Incomplete Blood Count Recovery (CRi) rate as defined by 2003 International Working Group (IWG) for AML.
Overall Response Rate (ORR) | Up to 12 months
  Overall Response Rate is defined as CR + CRi + partial response (PR) as defined by 2003 IWG criteria for AML.
Relapse Free Survival (RFS) | Up to 18 months
  RFS is defined as time interval between achievement of CR to time of relapse.
Overall Survival (OS) | Up to 12 months
  OS defined as time interval from time of enrollment onto the clinical trial to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Zhuoer Xie, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States